CLINICAL TRIAL: NCT03473873
Title: Is Good Muscle Function a Protective Factor for Early Features of Knee Osteoarthritis After Anterior Cruciate Ligament Injury (SHIELD)? A Prospective Cohort Study
Brief Title: Protective Role of Muscle Function for Early Features of Knee Osteoarthritis After Anterior Cruciate Ligament Injury
Acronym: SHIELD
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/319
Record Dates: First submitted 2018-03-09; First posted 2018-03-22 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis; Anterior Cruciate Ligament Injury; Osteoarthritis, Knee; Muscle Weakness
MeSH Terms: conditions — Osteoarthritis, Knee; Anterior Cruciate Ligament Injuries; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SHIELD: Patients with anterior cruciate ligament injury
  Interventions: Other: Measures of muscle function

INTERVENTIONS:
Other: Measures of muscle function — The participants will be assessed with various measures of muscle function at baseline and at follow up including: Isokinetic knee muscle strength, Isometric strength of trunk and lower extremity, single-leg hop for distance (SLHD), side hop, postural orientation errors (single leg-squat, stair descending, forward lunge, SLHD), hip and ankle range of motion, and muscular activation patterns.

SUMMARY:
In this longitudinal prospective cohort study including young people with anterior cruciate ligament reconstruction (ACLR), the aims are to 1) study the association between different measures of muscle function and early future of knee osteoarthritis (OA) assessed as patient-reported pain, 2) explore potential associations between muscle function and features indicative of early radiographic OA measured with MRI, and early detection of OA in biomarker profiles, respectively, 3) monitor the patients' functional status, and early OA development over time and 4) investigate the prevalence of early knee OA in individuals 1 and 3 years post ACLR, respectively, compared to non-injured controls.The main hypothesis is that knee extensor weakness predicts future symptomatic OA of the knee (KOOS pain).

DETAILED DESCRIPTION:
This is a longitudinal, prospective, cohort study. The reporting will adhere to the STROBE guidelines. Approximately 100 patients 12 months (range 10 - 16 months) after anterior cruciate ligament reconstruction (ACLR) will be recruited from Skåne University Hospital, Sweden and Ullevål Hospital, Oslo, Norway. The majority of the patients (approx. 80 %) will be recruited in Sweden. As a sample of convenience, 20 age- and sex-matched non-knee injured individuals will be recruited among students in Lund, Sweden.

A research coordinator at each site will determine eligibility for the study, based on pre-specified inclusion and exclusion criteria. Patients will be provided with written and oral information about the study. Patients who accept to participate will be assessed with various measures of muscle function, patient-reported outcomes, MRI, and blood samples for biomarker analyses, at baseline (1 year after ACLR) and 2 years later (3 years after ACLR).

For descriptive purposes, the mean difference (95% CI), or median (quartiles), between baseline and follow-up assessments will be used as appropriate. Separate linear regression model will be used to elucidate the influence of change in each muscle function variable on change in primary, secondary and exploratory outcomes (biomarkers), adjusted for baseline values. Separate linear regression models will also be used to elucidate the influence of demographic factors on change in muscle function, self-reported outcomes, and early OA. Assuming a clinically relevant correlation of 0.30 between knee extension strength and self-reported pain, 84 patients are needed with 80% power at the 5% significance level. Based on this calculation, 100 patients will be included, including an approximate drop-out of 15%. For explorative purposes, an analysis of covariance (ANCOVA) will be used to investigate differences in the presence of early knee OA between the 100 patients with ACLR and twenty sex and age matched non-injured individuals, adjusting for activity level.

ELIGIBILITY:
Inclusion Criteria patients:

* One year after ACL reconstruction (ACLR)
* With or without associated injuries to other structures of the knee (e.g., collateral ligament(s), meniscal injury)
* Age 18-35 years

Inclusion Criteria controls:

* Age 18-35 years
* No previous injuriy or surgery to either knee

Exclusion Criteria:

* Less than 10 months after ACLR
* More than 16 months after ACLR
* Injury or surgery to other knee (e.g., ACL, meniscal)
* Previous knee surgery index knee
* Previous serious knee injury index knee resulting in pain, swelling, and/or requiring inpatient or outpatient health care (e.g., ACLR, meniscus, patella luxation)
* Diseases or disorders overriding the knee condition (e.g., neurological disease)
* Contraindications for MRI
* Not understanding the languages of interest (any Scandinavian language or English)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited from the Department of Orthopedics, Skåne University Hospital, Sweden and the Department of Orthopedics, Ullevål Hospital, Oslo, Norway. The majority of patients (approx. 80%) will be included in Sweden.
  Non-injured controls will be recruited among students at Lund University, Lund, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Patient-reported pain | Change from baseline to 2-year follow up
  Knee Osteoarthritis Outcome Score (KOOS) subscale pain

SECONDARY OUTCOMES:
Compositional MRI (T2 relaxation time and 3DPD) | Change from baseline to 2-year follow up
  Compositional MRI, a proxy for early morphological degeneration of joint structures. Quantitative morphology of cartilage quality will be made using T2 mapping, to measure collagen orientation changes within the cartilage, and bone shape (3DPD)

OTHER OUTCOMES:
Biomarkers | Change from baseline to 2-year follow up
  Blood samples of venous blood will be collected to assess molecular biomarkers of cartilage turnover in serum. Specific biomarkers including, but not limited to, Cartilage oligomeric matrix protein (COMP), will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ageberg, PhD, Principal Investigator — Department of Health Sciences, Lund University, PO Box 157, 221 00 Lund, Sweden; May Arna Risberg, PhD, Principal Investigator — Oslo University Hospital, Division of Orthopedic Surgery, PO.Box 4956 Nydalen, 0424 Oslo, Norway
Locations (2):
- May Arna Risberg, Oslo, Norway
- Eva Ageberg, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided